CLINICAL TRIAL: NCT06777615
Title: Electronic Archive of Patients With Congenital Heart Disease and Diagnosis of Infective Endocarditis
Acronym: IE-CHD
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: IE-CHD
Record Dates: First submitted 2024-12-30; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Congenital Heart Disease (CHD); Infective Endocarditis (IE)
MeSH Terms: conditions — Heart Defects, Congenital; Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study is to create an electronic archive in which to census all newly diagnosed or already diagnosed cases of infective endocarditis and congenital heart disease after 01 January 2022 at the IRCCS AOU Bologna Pediatric and Developmental Age Cardiology Center so that be able to describe the clinical and echocardiographic features in patients with congenital heart disease and infective endocarditis in this population in order to be able to define new diagnostic/epidemiological hypotheses and the identification of predictive factors of adverse outcome (death, re-intervention, re-hospitalization) in patients with congenital heart disease and EI.

DETAILED DESCRIPTION:
It is well known in the literature that in patients with congenital heart disease, the risk of developing infective endocarditis (IE) is higher than in the general population with significant variation according to the underlying heart disease.It is essential to identify patients with congenital heart disease at higher risk of developing infective endocarditis and its related complications.Therefore, it is necessary to study the case history of patients with infective endocarditis and heart disease congenital heart disease (analysis of clinical-instrumental data, medical history, comorbidities, the cardiovascular adverse events and population mortality). The objective of the study is to create an electronic archive in which to census all newly diagnosed or already diagnosed cases of infective endocarditis and congenital heart disease after 01 January 2022 at the IRCCS AOU Bologna Pediatric and Developmental Age Cardiology Center so that be able to describe the clinical and echocardiographic features in patients with congenital heart disease and infective endocarditis in this population in order to be able to define new diagnostic/epidemiological hypotheses and the identification of predictive factors of adverse outcome (death, re-intervention, re-hospitalization) in patients with congenital heart disease and EI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital heart disease and established diagnosis of infective endocarditis referred to the UO Cardiology and Pediatric Cardiac Surgery Dell'IRCCS AOU of Bologna from 01/01/2000 until to approval (retrospective phase) and from approval until at least 31/12/2027 (prospective phase)
* Obtaining informed consent for participation in the study

Exclusion Criteria:

* no one

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with bacterial endocarditis and congenital heart disease will be considered, referred to our center from 01 January 2000 and until at least 31 December 2027 going to include, according to a preliminary analysis, a cohort of about 30 patients for the two phases in the above period.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify predictive factors of adverse outcome (death, re-intervention, re-hospitalization) in patients with congenital hea | Through study completion, an average of 5 years
  mortality, and related cause, re-hospitalization following diagnosis of EI (infective endocarditis).

CONTACTS AND LOCATIONS:
Overall Officials: Ylenia Bartolacelli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No